CLINICAL TRIAL: NCT05850858
Title: Platelets to Lymphocytes Ratio and Monocytes to Lymphocytes Ratio as Predictors of Response to Treatment in Cirrhotic Patients With Spontaneous Bacterial Peritonitis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mohamed Hamed Mohamed, Platelets to Lymphocytes Ratio and Monocytes to Lymphocytes Ratio as Predictors of Response to Treatment in Cirrhotic Patients with Spontaneous Bacterial Peritonitis, Sohag University
Other Study IDs: Soh-Med-23-04-11-MS
Record Dates: First submitted 2023-04-30; First posted 2023-05-09 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-04

CONDITIONS: Cirrhotic Patients With Spontaneous Bacterial Peritonitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cirrhotic Patients with Spontaneous Bacterial Peritonitis
  Interventions: Diagnostic Test: ascetic fluid study
- patient liver cirrhosis (child B,C)
- normal individuals

INTERVENTIONS:
Diagnostic Test: ascetic fluid study — ascetic fluid study parameter in diagnosis of spontaneous bacterial peritpnitis
  Groups: Cirrhotic Patients with Spontaneous Bacterial Peritonitis

SUMMARY:
Spontaneous bacterial peritonitis (SBP) is a serious complication of ascites that can lead to death and can be described as an acute infection of ascites without any certain source of infection SBP is considered the most common infection in cirrhotic patients with ascites. SBP is diagnosed by the presence of ≥250 polymorphonuclear leukocyte (PMNL)/mm3 in the ascetic fluid in absence of surgical and treatable causes of intra-abdominal infections .

SBP has many pictures of clinical presentation SBP can be asymptomatic and patients pass unnoticed or can discovered accidentally may have local symptoms and signs of peritonitis such as abdominal pain, and tachypnea or may present with signs of deteriorated liver function in form of gastrointestinal bleeding, shock and renal failure An increasing amount of studies have demonstrated that peripheral blood neutrophil-to-lymphocyte ratio (NLR), monocyte-to-lymphocyte ratio (MLR), platelet-to-lymphocyte ratio (PLR) are indicators of systematic inflammatory response and are widely investigated as useful predictors of the clinical outcomes in various diseases .

ELIGIBILITY:
Inclusion Criteria:

* Cirrhotic patient with ascites.
* Un treated SBP

Exclusion Criteria:

* Ascites without cirrhosis (malignant ascites, chylous ascites, etc…).
* Tuberculous peritonitis.
* Secondary bacterial peritonitis due to any surgical cause.
* Sepsis rather than SBP.
* Patients with unrelated infections e.g. skin, chest infection, etc.
* Patients started treatment of SBP.
* Patients on prophylactic antibiotics for recurrent SBP prevention .
* Patients declining to provide informed consent.
* Patients with hepatocellular carcinoma on top of cirrhosis.
* Patients with other malignancy or any immunological disease

Ages: 15 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Asses the value of blood platelets to lymphocytes ratio and monocytes to lymphocytes ratio as predictors of response for the treatment of spontaneous bacterial peritonitis in cirrhotic patients.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-04-19 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Platelets to Lymphocytes Ratio and Monocytes to Lymphocytes Ratio as Predictors of Response to Treatment in Cirrhotic Patients with Spontaneous Bacterial Peritonitis | 19/4/2023 - 30/4/2024
  Spontaneous bacterial peritonitis (SBP) is a serious complication of ascites that can lead to death and can be described as an acute infection of ascites without any certain source of infection SBP is considered the most common infection in cirrhotic patients with ascites. SBP is diagnosed by the presence of ≥250 polymorphonuclear leukocyte (PMNL)/mm3 in the ascetic fluid in absence of surgical and treatable causes of intra-abdominal infections SBP has many pictures of clinical presentation SBP can be asymptomatic and patients pass unnoticed or can discovered accidentally may have local symptoms and signs of peritonitis such as abdominal pain, and tachypnea or may present with signs of deteriorated liver function in form of gastrointestinal bleeding, shock and renal failure

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

REFERENCES:
- [Background] Song DS. [Spontaneous Bacterial Peritonitis]. Korean J Gastroenterol. 2018 Aug 25;72(2):56-63. doi: 10.4166/kjg.2018.72.2.56. Korean. PMID 30145857
- [Background] Abdel Hammed MR, El-Amien HA, Asham MN, Elgendy SG. Can platelets indices and blood neutrophil to lymphocyte ratio be used as predictors for diagnosis of spontaneous bacterial peritonitis in decompensated post hepatitis liver cirrhosis? Egypt J Immunol. 2022 Oct;29(4):12-24. PMID 36197150
- [Background] Chen TM, Lin CC, Huang PT, Wen CF. Neutrophil-to-lymphocyte ratio associated with mortality in early hepatocellular carcinoma patients after radiofrequency ablation. J Gastroenterol Hepatol. 2012 Mar;27(3):553-61. doi: 10.1111/j.1440-1746.2011.06910.x. PMID 21913982